CLINICAL TRIAL: NCT06705582
Title: A Dietary Intervention Study to Evaluate the Efficacy of Fortified Bread in Preventing Low Vitamin D Status Among Older Adults During Wintertime in Ireland
Brief Title: OASIS Study: Vitamin D Deficiency Prevention Among Older Adults in Ireland
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Mairead Kiely PhD, Professor, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OASIS
Record Dates: First submitted 2024-11-15; First posted 2024-11-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fortified bread (Experimental): Intervention group will be supplied with fortified bread
  Interventions: Other: Fortified Bread
- Unfortified bread (Placebo Comparator): Control arm will receive unfortified bread and dietary advice to incorporate fortified foods that are commonly available on the market in their diet.
  Interventions: Other: Unfortified bread

INTERVENTIONS:
Other: Fortified Bread — Intervention group will be supplied with fortified bread delivering 10 -15 μg (400-600 IU) vitamin D3 in a daily portion and will receive dietary advice to incorporate fortified foods that are commonly available on the market in their diet.
  Arms: Fortified bread
Other: Unfortified bread — Placebo control group will be supplied with unfortified bread and will receive dietary advice to incorporate fortified foods that are commonly available on the market in their diet.
  Arms: Unfortified bread

SUMMARY:
Vitamin D deficiency is common. It is caused by limited sun availability together with a low supply of vitamin D in the food system. There is a high prevalence of low vitamin D status around the world. In Ireland, our relatively northern latitude and prevailing weather mean that UVB availability for skin synthesis of vitamin D is limited in this country and our population relies on the dietary supply of vitamin D to prevent deficiency. Thus, the endemic Irish problem of vitamin D malnutrition is due to the lack of vitamin D in our food system. Dietary guidelines cannot address this issue because foods naturally rich in vitamin D are very few and infrequently consumed.

The OASIS study will test the hypothesis that a vitamin D-fortified bread as part of a healthy diet that includes vitamin D-fortified foods is effective in preventing low vitamin D status during winter, and safe for older adults to consume.

DETAILED DESCRIPTION:
This randomised controlled dietary intervention study aims to recruit 200 older adults (>65 years) who will be randomised to receive vitamin D-fortified bread and advice to consume additional commercially available fortified foods (Treatment group) or identical unfortified bread and advice to consume additional commercially available fortified foods (Control group). The outcome of the study is to test whether increasing vitamin D intake through food (Treatment group) is sufficient to prevent wintertime vitamin D deficiency (measured using serum concentrations of 25-hydroxyvitamin D <30 nmol/L) in comparison with the Control group.

The target vitamin D intake for the treatment group in this study is >15-20 μg/day vitamin D. This will maintain serum concentrations of 25-hydroxyvitamin D (25(OH)D) (the biomarker of vitamin D status) > 30 nmol/L, the clinical deficiency threshold to prevent metabolic bone disease, in over 90% of participants. At this vitamin D intake level, about 80% of participants will have a 25(OH)D concentration > 50 nmol/L, the personal intake target in the US and EU.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Be an adult ≥65 years.
3. Willing to consume bread provided and have storage capacity for frozen bread.
4. Be in good general health.
5. Be willing to follow the assigned diet for 10 weeks and attend the required appointments.

   -

Exclusion Criteria:

Regularly consume a single high dose vitamin D supplement (>10µg/d /400 IU equivalent).

2. Exposure to factors that may influence vitamin D status, such as winter sun holiday, tanning bed usage.

3. Are following a medically prescribed diet. 4. Have a diagnosis of an acute or chronic medical condition that in the opinion of the investigator would interfere with the outcomes of the study such as Coeliac disease, Inflammatory Bowel Disease, liver disease, renal disease, pancreatic disease or gastric disease.

5. Have a history of active cancer or a diagnosis of cancer within the past 5 years.

6. Are taking certain medications that can impact vitamin D status, such as glucocorticoids.

8. Have regular excessive alcohol intake (≥28 units per week). 9. Have a known food allergy. 10. Are participating in another research study with an intervention or other lifestyle programme that would interfere with the outcomes of the study.

11. Are unable to read, write, or understand English.

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of 25-hydroxyvitamin D (25(OH)D) | 10 weeks
  Comparison of the number of participants with low vitamin D status (e.g. <30 nmol/L and < 50 nmol/L serum 25(OH)D) between treatment and placebo groups

SECONDARY OUTCOMES:
Vitamin D intakes | 10 weeks
  Comparison of prevalence of inadequate vitamin D intakes relative to North American and European dietary recommendations
Serum concentrations of albumin-corrected serum calcium concentrations as a safety measure | 10 weeks
  Comparison of albumin-corrected serum calcium concentrations < 2.6 mmol/L between treatment and placebo control groups
Circulating biomarkers of metabolic health status | 10 weeks
  Comparison of circulating biomarkers of metabolic health status and metabolomic markers between active and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Mairead E Kiely, PhD, Principal Investigator — University College Cork
Locations (2):
- Ireland (2):
  - Human Nutrition Studies Unit, School of Food and Nutritional Sciences, Cork, Cork
  - UCD Institute of Food and Health, Dublin, Dublin

IPD SHARING:
Plan to Share IPD: No
Please contact m.kiely@ucc.ie for any queries related to data access